CLINICAL TRIAL: NCT03265093
Title: Current Approach in the Treatment of Lichen Planus: Injectable Platelet Rich Fibrin ((İ-PRF)
Brief Title: Use of Injectable Platelet Rich Fibrin in Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EbSAGLAM2
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Lichen Planus
Keywords: Pain Measurement; Platelet Activation; Quality of Life
MeSH Terms: conditions — Lichen Planus | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Blinded, Parallel group, randomized controlled trial
Who Masked: Investigator
Masking Description: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental; Corticosteroid (Active Comparator): Intralesional corticosteroid administration
  Interventions: Drug: Corticosteroid
- Experimental; Injectable Platelet rich fibrin (Experimental): Injectable Platelet rich fibrin
  Interventions: Other: Platelet Rich Fibrin Injection

INTERVENTIONS:
Other: Platelet Rich Fibrin Injection — Venous blood will be taken from the patient every session and I-PRF will be created in the centrifuge. I- prf will be injected on one side and corticosteroid will be injected on the other side in patients with bilateral oral lichen planus. Once a week in the first month after treatment and one time at the end of the second month, the patient will be called to the control.
  Arms: Experimental; Injectable Platelet rich fibrin
Drug: Corticosteroid — Corticosteroid injection
  Arms: experimental; Corticosteroid

SUMMARY:
Platelet Rich Fibrine (PRF), which promotes wound healing by supporting angiogenesis, immunity and epithelial proliferation phases. over a decade has since past since PRF was developed and many clinicians now point to the potential use of a liquid version of PRF. a liquid injectable-platelet-rich fibrin (i-PRF) was developed by modifying spin centrifugation forces. At lower centrifugation speeds and by utilizing non-glass centrifugation tubes, the fibrin coagulation could be slowed down at early time points thus generating an injectable PRF. Much like traditional PRF, i-PRF contains an increase in leukocyte number and is further able to stimulate growth factor release.

Lichen planus is a common chronic mucocutaneous inflammatory disorder which generally affect s middle aged adults. Therapeutic methods including topical and systemic corticosteroids for the treatment of oral lichen planus (OLP) are suggested. However, long

-term use of corticosteroids may be associated with local and systemic complications, and moreover, some patients may not be responsive.

The investigators aimed to apply a treatment of autogenous origin (including no foreign products), considering the side effects of our corticosteroids. The study was designed as a split mouth.

The investigators planned to administer I-PRF to one side and intralesional corticosteroid therapy to the other side at patients with bilateral atrophic / erosive oral lichen planus lesions

DETAILED DESCRIPTION:
Lichen planus diagnosis will be made histopathologically. Intraoral photographs and measurements will be taken at the beginning of the treatment and 2 months after the treatment is finished.

ELIGIBILITY:
Inclusion Criteria:

1. Oral erosive lesions were diagnosed according to Andreasen classification.
2. Histological confirmation of erosive OLP according to the World Health Organization's clinicopathological diagnostic criteria for OLP.
3. No previous treatment of oral lichen planus at least 3 months.
4. Willingness and ability to complete the present clinical trial.
5. Patients of ages above 18 years old without skin involvement.

Exclusion Criteria:

1. Histological signs of dysplasia.
2. Using drugs associated with lichenoid reaction.
3. Pregnant, lactating and smoker patients.
4. Patient with systemic diseases such as diabetes mellitus, immunodysfunction, hematological and hepatological patients or had photosensitivity history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 6 months
  Patients were asked to grade the severity of their symptoms in numbers from 1(very mild pain) to 100 (very sever pain) on the visual analog scale in each visit.
Thongprasom sign scoring system | 6 months
  The lesions were evaluated according to Thongprasom sign scoring system
Oral Health- Related Quality of Life index (OHIP-14) | 6 months
  Patients were asked to grade the Oral Health- Related Quality of Life index

SECONDARY OUTCOMES:
Oral Hygiene Index | 6 months
  Oral Hygiene Index were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Sağlam, PhD, Study Chair — Bezmialem Vakif University; Mustafa Tunalı, Assoc. prof., Study Director — Bezmialem VakifUniversity; Tuğba Ünver, PhD, Principal Investigator — Bezmialem Vakif University; Zeliha Betül Özsağır, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Ebru SAĞLAM, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided